CLINICAL TRIAL: NCT03855358
Title: A Phase Ib Study of TQB2450 Injection and Anlotinib Hydrochloride Capsules to Treat Triple Negative Breast Cancer (TNBC)
Brief Title: A Study of TQB2450 Injection and Anlotinib Hydrochloride Capsules to Treat Triple Negative Breast Cancer (TNBC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-07
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-02

CONDITIONS: Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 Injection and Anlotinib Hydrochioride Capsules (Experimental)
  Interventions: Drug: TQB2450 Injection and Anlotinib Hydrochioride Capsules

INTERVENTIONS:
Drug: TQB2450 Injection and Anlotinib Hydrochioride Capsules — TQB2450 1200mg intravenously (IV) every-3-weeks (Q3W) and Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PD-L1 inhibitorin in combination with Anlotinib treatment for patients with triple receptor negative breast cancer treated after failure of standard therapy (including Anthracyclines and/or Taxanes).

ELIGIBILITY:
Inclusion Criteria:

- 1、18 and 75 years old; ECOG physical condition: 0 - 1 points; expected survival time more than 3 months。 2、Histological or cytological diagnosis of relapsed/metastatic triple receptor negative breast cancer (TNBC).TNBC is defined negatively expression of estrogen(ER), progesterone(PR) and human epidermal receptor-2(HER2).If there is a pathology report of the metastasis, take the histopathology of the metastases as standard. Negative of ER and PR is defined as expression of ER,PR<1% of the tumor cells by immunohistochemistry (IHC). HER2-negative is defined as a score of 0 and 1+ by IHC, or IHC 2+ & fluorescent in situ hybridization (FISH)negative. If the ER2 test result is 0 or 1+ by IHC, FISH detection is optional, but the result must be negative.

3、Patients had at least one measurable lesion (RECIST 1.1); 4、Participants has received prior anthracyclines and/or taxanes in first-line therapy. Disease progressed after latest chemotherapy. For adjuvant therapy/neoadjuvant therapy, disease relapse or progression during treatment or within 6 months after treatment is considered as failure of standard therapy.

5、Subject must have adequate organ functions and meet requirements on laboratory values.：Count of Blood Cells:hemoglobin content(HB)≥80g/L（No blood transfusion was performed within 14 days）； absolute neutrophil count (ANC) ≥ 1.5 × 10^9 / L; platelet count (PLT) ≥ 75 × 10^9 / L;; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN，with the exception of patients with hepatic metastases (ALT and AST ≤ 5 × ULN) , Biochemical examination: serum total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN), with the exception of patients with Gilbert's syndrome(TBIL≤3×ULN） ; serum creatinine (Cr) ≤ 1.5 × ULN or Creatinine clearance rate>50 μmol/L;Blood coagulation function:Prothrombin time(PT)≤1.5×ULN、International standardized ratio(INR)≤1.5×ULN、Activation partial thrombin time(APTT)≤1.5×ULN、Prothrombin time≤1.5×ULN；Doppler ultrasound evaluation：Left ventricular ejection fraction（LVEF)≥50%×ULN. 6、Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug and should agree to use an adequate method of contraception starting with the first dose of study therapy through 8 weeks after the last dose of study therapy.Men enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 8 weeks after the last dose of study therapy； 7、Subject has voluntarily agreed to participate by giving written informed consent.

Exclusion Criteria:

1. Patients previously treated with vegfr-targeted inhibitor drugs, including anrotinib hydrochloride capsules, or with other pd-1 / pd-l1 / ctla-4 antibodies or other immunotherapy for pd-1 / pd-l1 / ctla-41;
2. the people who get other monoclonal antibodies have severe hypersensitivity ;
3. Present or along with other malignancies within 5 years.Except for carcinoma in situ of the cervix, intramucosal carcinoma of the gastrointestinal tract, breast cancer and non-melanoma skin cancer and superficial bladder tumor[Ta,Tis,Ti];
4. Has any active autoimmune disease or a history of autoimmune disease (as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis;Subjects with asthma requiring medical intervention with bronchodilators were excluded）.However, the following patients were allowed to be enrolled: vitiligo, psoriasis, hair loss without systemic treatment, well-controlled type I diabetes, and hypothyroidism with normal thyroid function after alternative treatment；
5. Immunosuppressive therapy (>10mg/ day prednisone or other therapeutic hormones) with systemic or absorbable topical hormone therapy is required and replacement therapy for hypothyroidism with normal thyroid function is required within 2 weeks of the first dose；
6. Patients with multiple factors affecting oral medication (such as inability to swallow, gastrointestinal tract resection, chronic diarrhea, and intestinal obstruction)；
7. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage；
8. Patients with any signs of bleeding or a history of physical illness, regardless of severity;Patients with any bleeding or bleeding event more than CTCAE 3 level within 4 weeks before the first administration;Or the presence of unhealed wounds, fractures, gastric and duodenal active ulcers, ulcerative colitis and other gastrointestinal diseases or the presence of active bleeding in unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the researchers;
9. Patients have uncontrollable symptoms of brain metastasis, spinal cord compression, cancerous meningitis, or diseases found in CT or MRI during screening within 8 weeks before the first administration;
10. four weeks before the start of study treatment has been approved or in the research of anti-tumor treatment, including but not limited to, surgery, radiation therapy, chemotherapy, biological target therapy, interventional therapy, immune therapy and anti-tumor Chinese medicine therapy (to be based on the instroction of Chinese traditional medicine, after 2 weeks elution phase can also be set)and so on (note: people who oral targeted drug is less than five drugs half-life;Or oral fluorouracil drugs less than 14 days, mitomycin C and nitroso urea less than 6 weeks;Patients with adverse events (except hair loss) caused by previous treatment did not recover to a level less than or less than CTCAE 1；
11. Any patient with any serious and / or non controlled disease，including:a)The blood pressure control is not ideal (more than 150 mmHg systolic blood pressure，diastolic blood pressure greater than 90 mmHg) patients；b)Unstable angina, myocardial infarction, grade 2 or more than grade 2 congestive heart failure within 6 months after first administration, or arrhythmia requiring treatment (including QTc more than 480ms)；c)The activity or failed to control severe infection (more than II level of AE CTC infection)；d)Carriers of hepatitis b virus with a known clinical history of liver disease, including viral hepatitis, must be excluded from active HBV infection, i.e., HBV DNA positive (>1 10^4 copy /mL or >2000IU/mL);Known hepatitis c virus infection (HCV) and HCV RNA positive (>1 x 10^3 copy /mL), or other decompensated liver disease, chronic hepatitis requires antiviral treatment; e)HIV test positive; f)The poor diabetes control (fasting blood glucose (FBG)more than CTCAE 2)；
12. Inoculated with preventive vaccine or attenuated vaccine within 4 weeks after the first dose;
13. according to the judgment of the researcher, the subject may have other factors that may cause the termination of the study. For example, other serious diseases (including mental diseases) need to be treated together, there are serious laboratory examination abnormalities, accompanied by family or social factors, which may affect the safety of the subject or the collection of data and samples。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | Up to 72 weeks
  Overall Response Rate (ORR) defined as the proportion of subjects who achieves a best response of CR or PR, assessed by IRC per the Lugano Classification

SECONDARY OUTCOMES:
Complete Response (CR) | Up to 96 weeks
  Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis).
Overall Survival (OS) | Up to 96 weeks
  From the first dose of TQB2450 to the date of death
Duration of Response (DCR) | Up to 96 weeks
  The percentage of cases with remission (PR+CR) and stable disease (SD) after treatment in the evaluable cases

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China